CLINICAL TRIAL: NCT07238569
Title: Multicenter, Prospective Phase III Clinical Trial of EBV-DNA-Guided Adaptive Immunotherapy for Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Phase III Trial of EBV-DNA-Guided Adaptive Immunotherapy for Advanced Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-346-FLK
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Nasopharyngeal Cancinoma (NPC); Nasopharangeal Cancer
Keywords: adebrelimab; PD-L1 antibody; chemoradiotherapy; capecitabine
MeSH Terms: interventions — Immune Checkpoint Inhibitors; Cisplatin; Radiotherapy, Intensity-Modulated; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- adebrelimab plus capecitabine (Experimental): Patients will receive definitive intensity-modulated radiotherapy (IMRT) of 6996cGy in 33 fractions. Concurrent cisplatin of 100mg/m2 will be administered every 3 weeks for 2 cycles during IMRT. Subsequently, adjuvant therapy with adebrelimab (1200 mg, d1) will be initiated for a total of 5 cycles, and capecitabine will be administered at 650 mg/m² orally twice daily for one year.
  Interventions: Drug: Adebrelimab (PD-L1 inhibitor); Drug: Cisplatin (100mg/m2); Radiation: Intensity-modulated radiotherapy; Drug: Capecitabine
- adebrelimab (Active Comparator): Patients will receive definitive intensity-modulated radiotherapy (IMRT) of 6996cGy in 33 fractions. Concurrent cisplatin of 100mg/m2 will be administered every 3 weeks for 2 cycles during IMRT. Subsequently, adjuvant therapy with adebrelimab (1200 mg, d1) will be initiated for a total of 5 cycles.
  Interventions: Drug: Adebrelimab (PD-L1 inhibitor); Drug: Cisplatin (100mg/m2); Radiation: Intensity-modulated radiotherapy

INTERVENTIONS:
Drug: Adebrelimab (PD-L1 inhibitor) — Adebrelimab 1200mg will be given every 3 weeks for 5 cycles in adjuvant chemotherapy
Drug: Cisplatin (100mg/m2) — Induction cisplatin 80mg/m2, every 3 weeks for 3 cycles before radiation; Concurrent cisplatin 100mg/m2, every 3 weeks for 2 cycles during radiation
Radiation: Intensity-modulated radiotherapy — Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy will be given in 33 fractions.
Drug: Capecitabine — Capecitabine was administered at 650 mg/m² orally twice daily for one year.
  Arms: adebrelimab plus capecitabine

SUMMARY:
This trial evaluated the efficacy of two adjuvant regimens following identical induction and concurrent chemoradiotherapy (IC+CCRT) in locoregionally advanced nasopharyngeal carcinoma (LANPC) patients with persistent EBV DNA positivity or stable disease after three IC cycles. The control arm received adjuvant adebrelimab, while the experimental arm received adebrelimab plus capecitabine.

DETAILED DESCRIPTION:
This study will enroll patients with stage II-III LANPC (AJCC 9th edition, excluding T3N0-1). After three cycles of induction chemotherapy (gemcitabine, cisplatin, and adebrelimab), eligible patients with persistent EBV DNA or stable disease will be randomized 1:1. All patients will undergo CCRT followed by adjuvant therapy. The control arm will receive five cycles of adebrelimab. The experimental arm will receive five cycles of adebrelimab in combination with capecitabine, which will be administered for one year.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤65 years
2. Patients with histologically confirmed non-keratinizing nasopharyngeal carcinoma according to WHO criteria.
3. Eastern Cooperative Oncology Group performance score of 0-1.
4. Tumor staged as II-III disease (AJCC 9th edition), excluding T3N0-1.
5. Adequate marrow function: white blood cell count > 4 × 10⁹/L hemoglobin >90g/L and platelet count >100×10⁹/L
6. Adequate hepatic and renal function：

   * Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
   * Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) ≤2.5×ULN
   * Alkaline phosphatase ≤ 2.5 × ULN
   * clearance rate ≥ 60 ml/min
7. Other laboratory and clinical criteria

   * Normal thyroid function, serum amylase and lipase, pituitary hormone levels, inflammatory markers, cardiac enzyme tests and electrocardiogram (ECG)
   * For patients aged >50 years with a history of smoking, normal pulmonary function test (PFT) results are required
   * For patients with abnormal ECG findings or a prior history of cardiovascular disease (not meeting any exclusion criteria listed in Item 8), additional assessments including myocardial function evaluation and cardiac ultrasound (echocardiography) must be performed, with results within normal limits
8. Patients with persistent EBV DNA positivity or stable disease following 3 cycles of induction chemotherapy (gemcitabine, cisplatin, and adebrelimab).
9. Patients must be informed of the investigational nature of this study and give written informed consent, and be willing and able to comply with the study schedule, including follow-up visits, treatment procedures, laboratory testing, and other protocol-related requirements.
10. Women of childbearing potential (WOCBP) must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of study drug (e.g., condoms, physician-guided regular use of oral contraceptives).

Exclusion Criteria:

1. Disease progression after induction chemotherapy
2. Positive for hepatitis B surface antigen (HBsAg) with hepatitis B virus DNA >1×103 copies/mL, positive for anti-hepatitis C virus (HCV) antibody , positive for anti-hepatitis C virus (HCV) antibody
3. Positive for anti-HIV antibody or diagnosed with acquired immunodeficiency syndrome (AIDS).
4. Active pulmonary tuberculosis: Patients with a history of active tuberculosis within the past year should be excluded regardless of treatment status. Patients with a history of active pulmonary tuberculosis more than one year prior should also be excluded, unless they received confirmed and regular anti-tuberculosis treatment.
5. Active, known, or suspected autoimmune diseases, including but not limited to uveitis, colitis, hepatitis, hypophysitis, nephritis, vasculitis, systemic lupus erythematosus, hyperthyroidism, hypothyroidism, and asthma requiring bronchodilators. Type I diabetes, hypothyroidism treated with replacement therapy, and skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia) are allowed.
6. History of interstitial lung disease or pneumonia requiring oral or intravenous corticosteroids within the past year; use of vancomycin within the past month.
7. Ongoing chronic systemic corticosteroid therapy (equivalent to or greater than prednisone >10mg per day) or any other immunosuppressive therapy. Patients received inhale or topical corticosteroid are allowed.
8. Uncontrolled cardiac conditions, such as:

   * Heart failure with New York Heart Association (NYHA) classification ≥ Class II;
   * Unstable angina;
   * History of myocardial infarction within the past year;
   * Supraventricular or ventricular arrhythmias requiring treatment or intervention
9. Pregnant or breastfeeding women (pregnancy testing should be considered for women of childbearing potential with active sexual life)
10. History or presence of other malignancies, except for adequately treated non-melanoma skin cancer, carcinoma in situ of the cervix, and papillary thyroid carcinoma.
11. Known hypersensitivity to macromolecule protein products or any component of adebrelimab.
12. Active infections requiring systemic treatment within 1 week prior to enrollment.
13. Administration of live vaccines within 30 days prior to the first dose of adebrelimab.
14. Factors significantly affecting the absorption of oral drugs, such as inability to swallow, chronic diarrhea, or intestinal obstruction.
15. History of organ transplantation or hematopoietic stem cell transplantation.
16. Any other condition assessed by the investigator as potentially compromising patient safety or compliance, such as severe illnesses requiring urgent treatment (including psychiatric disorders), significantly abnormal laboratory values, or other psychological, familial, or social risk factors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2031-05-23 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival (FFS) | 3 year
  From date of randomization until the date of first documented locoregional recurrence, distant metastasis, or death from any cause, whichever occurred first, assessed up to 74 months

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  From date of randomization until the date of death from any cause, whichever came first, assessed up to 74 months
Distant metastasis-free survival (DMFS) | 3 years
  From date of randomization until the date of first documented distant metastasis, whichever occurred first, assessed up to 74 months.
Locoregional recurrence-free survival (LRRFS) | 3 years
  From date of randomization until the date of first documented locoregional recurrence, whichever occurred first, assessed up to 74 months.
Tumor response | the time of completion of induction chemotherapy, radiotherapy, and adjuvant immunotherapy; from the date of enrollment until the date of the last time that tumorimaging and assessment of disease has been done, assessed up to 74 weeks
  Evaluation of tumor response as CR, PR, SD, PD, NA by clinicians
Adverse events (AEs) and serious adverse events (SAEs) | 3 years
  Graded according to CTCAE V5.0.
Quality of life (QoL) | week 1, 6, 24, 60, 72
  The change of QoL from randomization to the start of radiotherapy, the end of radiotherapy, 13-16 weeks after radiotherapy, 2 years and 3 years after randomization. The EORTC QoL questionnaire-C30 (EORTC QLQ-C30）version 3.0 will be used. This questionnaire comprises 30 questions, 24 of which are aggregated into nine multi-question scales, that is, five functioning scales (e.g., physical), three symptom scales (e.g., fatigue) and one global health status scale. The remaining six single-question (e.g., dyspnoea) scales assess symptoms. These 15 scales will be scored according to the official Scoring Manual. For the functional scales and the global health status scale, a higher score represents a better level of functioning or quality of life. For the symptom scales, a higher score indicates a greater severity of symptoms.
Failure-free survival (FFS) within different subgroups | 3 years
  analyses for FFS will be performed within the following subgroups: Epstein-Barr virus (EBV) DNA (≤4000copies/ml vs. >4000copies/ml), different PD-L1 expression levels, age, gender, performance status, T category, N category, and stage.

OTHER OUTCOMES:
Correlation between pre-treatment PD-L1 expression level and FFS | 3 years
  Pre-treatment PD-L1 expression level of tumor cell is evaluated centrally by means of immunohistochemical testing.
Evaluate failure-free survival in the subgroup of plasma Epstein-Barr virus DNA level | 3 years
  Subgroup analysis

IPD SHARING:
Plan to Share IPD: No
Complete de-identified patient data set will be submitted onto an online platform.